CLINICAL TRIAL: NCT03762694
Title: The Effect of Acupuncture for Insomnia in Breast Cancer Patients Undergoing Chemotherapy: A Randomized, Wait-list Controlled Pilot Study
Brief Title: The Effect of Acupuncture for Insomnia in Breast Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor LAO Lixing, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 18-526
Record Dates: First submitted 2018-12-02; First posted 2018-12-04 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Insomnia, Secondary; Breast Cancer Female; Chemotherapy
Keywords: Acupuncture; Insomnia; Breast cancer; Chemotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (EA) and Auricular Acupuncture (AA) (Experimental): 12 sessions acupuncture treatment (EA+AA) will be given twice a week for 6 weeks after randomization.
  Interventions: Device: Acupuncture
- Wait-list control (No Intervention): No treatment except routine care will be given at the first 6 weeks, followed by 12 sessions treatment as Acupuncture group.

INTERVENTIONS:
Device: Acupuncture — Electroacupuncture (EA) and Auricular Acupuncture (AA)
  Arms: Electroacupuncture (EA) and Auricular Acupuncture (AA)

SUMMARY:
This pilot study is designed to determine whether acupuncture is a feasible, effective and safe method for alleviating insomnia among breast cancer patients undergoing chemotherapy as compared with a wait-list control.

DETAILED DESCRIPTION:
Hypothesis:

Acupuncture is a feasible, effective and safe method for alleviation of insomnia symptoms in breast cancer patients undergoing chemotherapy as compared with a wait-list control.

Objective:

To determine whether the insomnia condition in the acupuncture group is significantly improved when compared to the wait-list control group.

Design and strategy:

This is a randomized, wait-list controlled, assessor-blinded trial. 30 subjects will be recruited and randomized (in 1:1 ratio) to receive either acupuncture treatment or wait-list control. All patients in the 2 groups will receive routine Western medical care for symptom management.

Study instrument:

Insomnia Severity Index (ISI) will be employed as a primary outcome assessment.

Intervention:

In the treatment group, 12 sessions acupuncture treatment (electroacupuncture & auricular acupressure) will be given twice a week for 6 weeks after randomization. In the wait-list control group, no treatment except routine care will be given at the first 6 weeks, followed by 12 sessions treatment as treatment group.

Main outcome measures:

Primary outcome: ISI scores will be measured at week 0, 3, 6, 10, 14.

Secondary outcomes:

Pittsburgh Sleep Quality Index, Sleep diary, Actiwatch, Functional Assessment of Cancer Therapy-Breast Cancer, and adverse events will be documented and compared between groups.

Data analysis: The primary endpoint will be the continuous ISI score. For the primary analysis, if normality of the ISI or its transformation can be achieved, a two-sample t-test on the average ISI score will be performed to access the significance of the treatment effects; otherwise, a nonparametric approach will be taken.

Expected outcome: ISI score of the acupuncture group is expected to be significantly lower than wait-list control group after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between 18 and 75 years of age;
2. Diagnosis of stage (American Joint Committee on Cancer (AJCC) TNM) I-IV breast cancer;
3. Currently receiving chemotherapy, or have completed chemotherapy no more than 6 months;
4. Insomnia onset after the diagnosis of breast cancer;
5. Insomnia occurs at least 3 nights per week, and presents for at least 1 month, with fulfilment of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic criteria for brief insomnia disorder;
6. Insomnia severity as defined by an ISI score of no less than 10 in the past 2 weeks;
7. Expected survival time of more than 6 months;
8. Ability to understand the nature of the study and willingness to give informed consent;
9. Ability to provide responses during outcome measurement.

Exclusion Criteria:

1. Insomnia before the diagnosis of breast cancer;
2. Other sleep disorder (e.g., obstructive sleep apnoea);
3. Shift work or irregular sleep pattern;
4. Severe visual, hearing or language defects;
5. Severe hematological dysfunction (platelet count <60,000/μL, haemoglobin <8 g/dL or absolute neutrophil count <1000/μL);
6. With pacemakers or other electronic implants that could interfere with electroacupuncture;
7. History of acupuncture use in the previous 3 months;
8. Participation in other clinical trials with intervention within 3 months of the beginning of the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | week 0, 3, 6 (primary outcome), 10, 14

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | week 0, 3, 6, 10, 14
Sleep diary | week 0, 6
Actigraphy | week 0, 6
Functional Assessment of Cancer Therapy-Breast Cancer | week 0, 6, 10, 14
Adverse events | week 0 to week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Zhang J, Qin Z, So TH, Chen H, Lam WL, Yam LL, Yan Chan P, Lao L, Zhang ZJ. Electroacupuncture Plus Auricular Acupressure for Chemotherapy-Associated Insomnia in Breast Cancer Patients: A Pilot Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211019103. doi: 10.1177/15347354211019103. PMID 34036813